CLINICAL TRIAL: NCT04743570
Title: Effects of Peripherally Acting µ-opioid Receptor Antagonists on Acute Pancreatitis - An Investigator-initiated, Randomized, Placebo-controlled, Double-blind Clinical Trial
Brief Title: Effects of Peripherally Acting µ-opioid Receptor Antagonists on Acute Pancreatitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Asbjørn Mohr Drewes (Other)
Collaborators: Odense University Hospital (Other); Hvidovre University Hospital (Other); University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Sponsor-Investigator, Asbjørn Mohr Drewes, Professor, Chief Physician, MD, PhD, DMSc, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAMORA_AP, PAMORA-1; 2020-002313-18 (EudraCT Number); N-20200060 (Other: North Denmark Region Committee in Health Research Ethics)
Record Dates: First submitted 2021-01-28; First posted 2021-02-08 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo treatment (Placebo Comparator): Placebo consisting of Ringer's lactate in matched volume to active drug is added to 1000 mL Ringer's lactate solution and given as a continues infusion over 24 hours using an infusion pump.
  Interventions: Drug: Placebo treatment
- Methylnaltrexone treatment (Active Comparator): 0.15 mg/kg methylnaltrexone will be dissolved in 1000 mL Ringer's lactate solution and given as a continues infusion over 24 hours using an infusion pump.
  Interventions: Drug: Methylnaltrexone treatment

INTERVENTIONS:
Drug: Placebo treatment — Active drug/placebo is given for the first 5 days of admission.
  Arms: Placebo treatment
Drug: Methylnaltrexone treatment — Active drug/placebo is given for the first 5 days of admission.
  Arms: Methylnaltrexone treatment

SUMMARY:
This study will investigate the effect of peripheral acting opioid antagonist (PAMORA) on the disease course of patients with acute inflammation of the pancreas (acute pancreatitis). The study will be conducted by treating hospitalized patients with acute pancreatitis with a PAMORA (methylnaltrexone).

DETAILED DESCRIPTION:
In this study, the effects of peripheral acting µ-opioid receptor antagonists (PAMORA) on disease development and progression in patients with acute pancreatitis (AP) will be investigated. Patients with AP will be administered Methylnaltrexone (Relistor®) intravenously. This medication is defined as the investigational product. Relistor® is approved and sold on the Danish marked for treatment of opioid-induced constipation. This PAMORA have not previously been investigated in patients with pancreatitis. The dose regimes for this study will be according to label. It has previously been shown, in patients with opioid-induced obstipation and healthy subjects, that opioid antagonism incl. PAMORA treatment increases gut motility, relaxes gastrointestinal sphincters, increases the intestinal water content and improves the immune response, without affecting analgesia. The affinity of PAMORAs to the µ-opioid receptors is much stronger than opioid analgesics. Therefore, they as antagonists have the potential to counteract the harmful effects of opioids on the gut mucosa, bacterial translocation and inflammation despite the high levels of exogenous opioids present in patients with pancreatitis. PAMORAs do not cross the blood-brain barrier and consequently do not interfere with analgesia or other central effects of opioids.

We hypothesize that treatment with the PAMORA methylnaltrexone will antagonize the harmful effects of opioids without reducing analgesia in patients with AP and hence reduce disease severity and improve clinical outcomes. If successful, this sub-study will for the first time document the effects of a targeted pharmacotherapy in AP with the potential benefit of improved patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent before any study specific procedures
* Able to read and understand Danish
* Male or female age between 18 and 80 years
* The researcher believes that the participant understands what the study entails, is capable of following instructions, can attend when needed, and is expected to complete the study
* The investigator will ensure that fertile female participants have a negative pregnancy test before treatment initiation and use contraception during the study period. The following methods of contraception, if properly used, are generally considered reliable: oral contraceptives, patch contraceptives, injection contraceptives, vaginal contraceptive ring, intrauterine device, surgical sterilization (bilateral tubal ligation), vasectomized partner, double barrier (condom and pessary), or sexual abstinence. Methods of contraception will be documented in the source documents
* At least two of the following criteria need to be fulfilled to establish a diagnosis of AP (according to the revised Atlanta criteria (16)): i) abdominal pain consistent with AP (acute onset of a persistent, severe, epigastric pain often radiating to the back); ii) serum amylase activity at least three times greater than the upper limit of normal; and iii) characteristic findings of AP on diagnostic imaging
* Predicted moderate or severe AP based on 2 or more systemic inflammatory response syndrome criteria upon admission

Exclusion Criteria:

* Definitive chronic pancreatitis according to the M-ANNHEIM criteria
* Known allergy towards study medication
* Known or suspected major stenosis or perforation of the intestines
* Known or suspected abdominal cancer (incl. intestine, pancreas and the biliary tree)
* Pre-existing renal insufficiency (defined as habitual estimated glomerular filtration rate below 45)
* Severe pre-existing comorbidities (assessed by investigator upon inclusion)
* Severe non-pancreaticobiliary infections or sepsis caused by non-pancreaticobiliary disease
* Child-Pugh class B or C liver cirrhosis
* Females that are currently lactating

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2023-04-09 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Pancreatitis activity scoring system | 48 hours after randomization
  Difference in Pancreatitis activity scoring system (PASS) score between the methylnaltrexone group and the placebo group. The PASS-score is a weighted score of presence of organ failure, number of criterias of Systemic Inflammatory Response Syndrome fulfilled, abdominal pain (0-10), morphine equivalent dose (mg) and tolerance to solid food. Minimum value is 0 and higher score is equal to higher disease activity.
  Documentation for the PASS can be found on the following link: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5519418/

SECONDARY OUTCOMES:
Pancreatitis activity scoring system | 24 hours after randomization and every 24 hours untill end of study at day 5 (after 120 hours) and again at the day 14 follow-up visit
  Difference PASS scores between subgroups
Difference in assessments of circulating proinflammatory marker | 24 hours after randomization and every 24 hours untill end of study at day 5 (after 120 hours) and again at the day 14 follow-up visit
  C-Reactive Protein (mg/L)
Difference in assessments of circulating pro- and anti-inflammatory markers | 24 hours after randomization and every 24 hours untill end of study at day 5 (after 120 hours) and again at the day 14 follow-up visit
  Interleukin-6, Interleukin-8, Interleukin-18, Tumor necrosis factor alpha, Cluster of Differentiation 163 (serum) (all measured in pg/mL)
Intestinal permeability | From 48 to 72 hours after randomization
  Difference in intestinal permeability between subgroups using the oral polyethylene glycol 400/4000 test
Intestinal motility | 5 (+/- 1 day) after randomization
  Difference in intestinal motility assessed by means of gut/colon transit using a CT-based radiopaque marker method between subgroups
Pancreatic complications | Day 5 (+/- 1 day) after randomization
  Difference in pancreatic complications (e.g. edema, fluid collections and necrosis) assessed and quantified with contrast-enhanced CT
Pain intensity | 24 hours after randomization and every 24 hours untill end of study at day 5 (after 120 hours) and again at the day 14 follow-up visit
  Difference between subgroups in pain intensity measured with the questionaire "modified Brief Pain Inventory short form" on visual analogue scale from 0-10 (0 is no pain and 10 is worst pain).
Gut function (BSFS) | 24 hours after randomization and every 24 hours untill end of study at day 5 (after 120 hours) and again at the day 14 follow-up visit
  Difference between subgroups in gut function assessed by The Bristol Stool Form Scale for assessment of stool frequency as well as stool consistency (scale from 1-7, where 1 is firmeste and 7 is softest)
Gut function (GSRS) | 24 hours after randomization and every 24 hours untill end of study at day 5 (after 120 hours) and again at the day 14 follow-up visit
  Difference between subgroups in gut function assessed by Gastrointestinal Symptom Rating Scale which is a disease-specific instrument of 15 items combined into five symptom clusters depicting reflux, abdominal pain, indigestion, diarrhea and constipation. The GSRS has a seven-point graded Likert-type scale, where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
Quantification of analgesics | 24 hours after randomization and every 24 hours untill end of study at day 5 (after 120 hours) and again at the day 14 follow-up visit
  Difference between subgroups in given dose of analgesics (separated into opioids and non-opioids) based on name, administration route and dose
Use of nutritional support | 24 hours after randomization and every 24 hours untill end of study at day 5 (after 120 hours) and again at the day 14 follow-up visit
  Difference between subgroups in the use of nutritional support with registration of the used of either oral nutrition, enteral or parenteral nutrition.
Days of hospitalization | Observation period starts from day of randomization and ends after 12 months or on the day of discharge which ever comes first
  Difference between subgroups in days of hospitalization and days on intensive ward
Use of invasive treatment | Observation period starts from day of randomization and ends after 12 months or on the day of discharge whichever comes first
  Difference between subgroups in use of invasive treatment (e.g. use of drain or surgery) measured in type and frequency of use
Mortality | Observation period starts from day of randomization and ends after 12 months or on the day of discharge whichever comes first
  Difference between subgroups in mortality rate
Health resource utilization | Observation period starts from day of randomization and ends after 12 months or on the day of discharge whichever comes first
  Difference in health resource utilization (measured in frequency and type of health services used (e.g. blood sample, MRI etc.) that can be converted into danish currency for economic analyses) between subgroups based on service codes (all services have unique service codes stored digitally).
Disease severity | Observation period starts from day of randomization and ends after 12 months or on the day of discharge whichever comes first
  Disease severity classified by the revised Atlanta classification system in 3 levels; Mild, Moderate or Severe acute pancreatitis. (Mild acute pancreatitis, with no organ failure, local or systemic complications, Moderately severe acute pancreatitis is with presence of transient organ failure, local complications or exacerbation of co-morbid disease. Severe acute pancreatitis with persistent organ failure (>48 h).

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn M. Drewes, Professor, Study Chair — Mech-Sense, Department of Medical Gastroenterology, Aalborg Hospital
Locations (4):
- Denmark (4):
  - Mech-Sense, Department of Medical Gastroenterology, Aalborg University Hospital, Aalborg, Jutland
  - Digestive Disease Center K, Bispebjerg University Hospital, Bispebjerg
  - Gastrounit, Hvidovre University Hospital, Hvidovre
  - Odense Pancreas Center, Svendborg

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Knoph CS, Cook ME, Novovic S, Hansen MB, Mortensen MB, Nielsen LBJ, Hogsberg IM, Salomon C, Neergaard CEL, Aajwad AJ, Pandanaboyana S, Sorensen LS, Thorlacius-Ussing O, Frokjaer JB, Olesen SS, Drewes AM. No Effect of Methylnaltrexone on Acute Pancreatitis Severity: A Multicenter Randomized Controlled Trial. Am J Gastroenterol. 2024 Nov 1;119(11):2307-2316. doi: 10.14309/ajg.0000000000002904. Epub 2024 Jun 25. PMID 38916223
- [Derived] Knoph CS, Cook ME, Fjelsted CA, Novovic S, Mortensen MB, Nielsen LBJ, Hansen MB, Frokjaer JB, Olesen SS, Drewes AM. Effects of the peripherally acting mu-opioid receptor antagonist methylnaltrexone on acute pancreatitis severity: study protocol for a multicentre double-blind randomised placebo-controlled interventional trial, the PAMORA-AP trial. Trials. 2021 Dec 19;22(1):940. doi: 10.1186/s13063-021-05885-3. PMID 34924020

DOCUMENTS (2):
  • Study Protocol (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT04743570/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT04743570/SAP_001.pdf